CLINICAL TRIAL: NCT02158676
Title: Effect of Prebiotic and Synbiotic Supplementation on Inflammatory Markers, Metabolic Parameters and Nutritional Status After Roux-en-y Gastric Bypass.
Brief Title: Effect of Prebiotic and Synbiotic Supplementation in Individuals Undergoing Roux-en-y Gastric Bypass.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Santa Catarina (Other)
Responsible Party: Principal Investigator, Erasmo Benicio Santos de Moraes Trindade, Doctor in Tropical Diseases, Universidade Federal de Santa Catarina
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 96156587
Record Dates: First submitted 2014-06-02; First posted 2014-06-09 (Estimated); Last update posted 2017-04-14 (Actual); Status verified 2017-04

CONDITIONS: Obesity
Keywords: Roux-en-y gastric bypass; Inflammatory markers; Nutritional status; Fatty acids; Glucose; Prebiotic; Synbiotic
MeSH Terms: conditions — Obesity | interventions — Prebiotics; Synbiotics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Prebiotic (Experimental): 6 g/day of prebiotic (fructooligosaccharides) for 15 days.
  Interventions: Dietary Supplement: Prebiotic
- Synbiotic (Experimental): 6 g/day of synbiotic (fructooligosaccharides + Lactobacillus paracasei LPC-37 + Lactobacillus rhamnosus HN001 + Lactobacillus acidophilus NCFM + Bifidobacterium lactis HN019) for 15 days.
  Interventions: Dietary Supplement: Synbiotic
- Placebo (Placebo Comparator): 6 g/day of placebo (maltodextrin) for 15 days.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Prebiotic — Fructooligosaccharides
  Arms: Prebiotic
Dietary Supplement: Synbiotic — Fructooligosaccharides + Lactobacillus paracasei LPC-37 + Lactobacillus rhamnosus HN001 + Lactobacillus acidophilus NCFM + Bifidobacterium lactis HN019
  Arms: Synbiotic
Other: Placebo — Maltodextrin
  Arms: Placebo

SUMMARY:
The study will recruit patients submitted to bariatric surgery. Individuals will be supplemented with 6g/day of prebiotic or synbiotic or placebo (maltodextrin) for 15 days. Immunological, metabolic and anthropometric parameters will be assessed before and after the supplementation. Our hypothesis is that prebiotic or synbiotic supplementation modulate plasma concentrations of immunological and metabolic parameters and anthropometric measures of subjects undergoing gastric bypass Roux-Y.

DETAILED DESCRIPTION:
The study will recruit patients submitted to roux-en-y gastric bypass. Individuals that meet the inclusion criteria will be randomized by means of a computer program on three study groups: 1) Prebiotic group: Oral supplementation with 6g/day of prebiotic for 15 days. 2) Synbiotic group: Oral supplementation with 6g/day of synbiotic for 15 days. 3) Placebo group (control): Oral supplementation with 6g/day of placebo (maltodextrin) for 15 days. Will be assessed the effects of supplementation on the plasma cytokines, plasma lipopolysaccharide (bacterial endotoxin), plasma cellular fatty acid profile, metabolic parameters (lipid profile, glycemic status and insulin resistance) and nutritional status. Blood samples will be collected before the surgery and the supplementation will begin 30 days after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 years and less than 65 years
* Body mass index (BMI)> 40kg/m2 or> 35kg/m2 with at least one comorbidity
* Failure in the non-pharmacological and pharmacological treatment.

Exclusion Criteria:

* Significant intellectual limitations without adequate family support.
* Uncontrolled psychiatric disorder.
* Alcohol dependence and / or illicit drugs dependence.
* Current use of anti-inflammatory drugs and / or antibiotics and / or immunosuppressants
* Display intolerance prebiotics and / or probiotics and / or symbiotic
* Having made use of prebiotic and / or probiotic and / or symbiotic prior to the study period.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2013-10; Primary Completion 2014-05 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Change in IL-1 beta concentrations | Baseline (before surgery); Day 30 (after surgery, before supplementation); Day 45 (after surgery, after supplementation).
  Will be evaluated IL-1 beta plasma concentrations in baseline which corresponds to the day that the patient will undergo surgery, in 30 days after surgery (before supplementation) and in 45 days after surgery (after supplementation).
Change in IL-6 concentrations | Baseline (before surgery); Day 30 (after surgery, before supplementation); Day 45 (after surgery, after supplementation).
  Will be evaluated IL-6 beta plasma concentrations in baseline which corresponds to the day that the patient will undergo surgery, in 30 days after surgery (before supplementation) and in 45 days after surgery (after supplementation).
Change in TNF-alpha concentrations | Baseline (before surgery); Day 30 (after surgery, before supplementation); Day 45 (after surgery, after supplementation).
  Will be evaluated TNF-alpha plasma concentrations in baseline which corresponds to the day that the patient will undergo surgery, in 30 days after surgery (before supplementation) and in 45 days after surgery (after supplementation).

SECONDARY OUTCOMES:
Change in nutritional status | Baseline (before surgery); Day 30 (after surgery, before supplementation); Day 45 (after surgery, after supplementation).
  Will be assessed anthropometric measures: weight and height (baseline, 30 and 45 days after surgery) for the classification of nutritional status according to BMI
Change in risk of inflammatory and nutritional complications | Baseline (before surgery); Day 30 (after surgery, before supplementation); Day 45 (after surgery, after supplementation)
  Will be calculated the CRP/albumin ratio, as proposed by Correa et al (2002), using the cutoff points proposed by the same author for the classification of high, medium, decreased or no risk.
Change in fasting glucose concentrations | Baseline (before surgery); Day 30 (after surgery, before supplementation); Day 45 (after surgery, after supplementation).
  Will be assessed the plasma concentrations of fasting glucose in baseline which corresponds to the day that the patient will undergo surgery, in 30 days after surgery (before supplementation) and in 45 days after surgery (after supplementation).
Change in fasting insulin concentrations | Baseline (before surgery); Day 30 (after surgery, before supplementation); Day 45 (after surgery, after supplementation).
  Will be assessed the plasma concentrations of fasting insulin in baseline which corresponds to the day that the patient will undergo surgery, in 30 days after surgery (before supplementation) and in 45 days after surgery (after supplementation).
Change in HOMA-IR index | Baseline (before surgery); Day 30 (after surgery, before supplementation); Day 45 (after surgery, after supplementation).
  Will be assessed the HOMA-IR index in baseline which corresponds to the day that the patient will undergo surgery, in 30 days after surgery (before supplementation) and in 45 days after surgery (after supplementation).
Change in glycated hemoglobin | Baseline (before surgery); Day 30 (after surgery, before supplementation); Day 45 (after surgery, after supplementation).
  Will be evaluated glycated hemoglobin in baseline which corresponds to the day that the patient will undergo surgery, in 30 days after surgery (before supplementation) and in 45 days after surgery (after supplementation).
Change in lipid profile | Baseline (before surgery); Day 30 (after surgery, before supplementation); Day 45 (after surgery, after supplementation).
  Will be evaluated lipid profile in baseline which corresponds to the day that the patient will undergo surgery, in 30 days after surgery (before supplementation) and in 45 days after surgery (after supplementation).
Change in plasma monounsaturated fatty acids | Baseline (before surgery); Day 30 (after surgery, before supplementation); Day 45 (after surgery, after supplementation).
  Will be assessed the proportion (%) of plasma monounsaturated fatty acids
Change in plasma polyunsaturated fatty acids | Baseline (before surgery); Day 30 (after surgery, before supplementation); Day 45 (after surgery, after supplementation).
  Will be assessed the proportion (%) of plasma polyunsaturated fatty acids
Change in plasma saturated fatty acids | Baseline (before surgery); Day 30 (after surgery, before supplementation); Day 45 (after surgery, after supplementation).
  Will be assessed the proportion (%) of plasma saturated fatty acids

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Fernandes, Master's, Principal Investigator — Universidade Federal de Santa Catarina
Locations (1):
- Hospital Universitário Polydoro Ernani de São Thiago, Florianópolis, Santa Catarina, Brazil

REFERENCES:
- [Result] Fernandes R, Beserra BT, Mocellin MC, Kuntz MG, da Rosa JS, de Miranda RC, Schreiber CS, Frode TS, Nunes EA, Trindade EB. Effects of Prebiotic and Synbiotic Supplementation on Inflammatory Markers and Anthropometric Indices After Roux-en-Y Gastric Bypass: A Randomized, Triple-blind, Placebo-controlled Pilot Study. J Clin Gastroenterol. 2016 Mar;50(3):208-17. doi: 10.1097/MCG.0000000000000328. PMID 25909598
- See also: URL for full text article — http://journals.lww.com/jcge/pages/articleviewer.aspx?year=2016&issue=03000&article=00009&type=abstract